CLINICAL TRIAL: NCT07370012
Title: Evaluation Of The Effectiveness Of Prism Adaptation Therapy In Patients With Complex Regional Pain Syndrome (CRPS) Type I
Brief Title: Prism Adaptation Therapy for CRPS Type 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, AYŞE ELİF ŞEN AKALIN, Physical Medicine and Rehabilitation Specialist, Ankara Etlik City Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AEŞH-EK1-2023-590
Record Dates: First submitted 2026-01-19; First posted 2026-01-27 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Complex Regional Pain Syndrome I (CRPS I); Distal Radius Fracture; CRPS (Complex Regional Pain Syndromes); Neuropathic Pain
Keywords: Upper Extremity Rehabilitation; Budapest Criteria; Pain Management; Neuropathic Pain; Kinesiophobia; Quality of Life; Ultrasonography / Edema grading; Hand Function; Complex Regional Pain Syndrome I; Complex Regional Pain Syndrome; CRPS; Prism Adaptation Therapy; Prism Adaptation; Neglect; CRPS I; Reflex Sympathetic Dystrophy; Prism Goggles; Visuomotor Adaptation; Sensorimotor Training; Body Perception Disturbance; Neglect-like Symptoms; Distal Radius Fracture; Upper Limb; Wrist; RSD
MeSH Terms: conditions — Complex Regional Pain Syndromes; Wrist Fractures; Neuralgia; Agnosia; Kinesiophobia; Reflex Sympathetic Dystrophy

STUDY DESIGN:
Intervention Model Description: Participants were divided into two groups: one group received prism adaptation therapy, while the other underwent the identical protocol using sham goggles.
Who Masked: Participant
Masking Description: Participants wore either prismatic-lens goggles or neutral-lens goggles during the pointing protocol. Both interventions were described as potentially beneficial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prism Adaptation Therapy Group (Active Comparator): The prism adaptation therapy intervention group
  Interventions: Device: The Prism Adaptation Therapy Group
- Control Group (Placebo Comparator): The control group that will undergo the protocol using sham goggles
  Interventions: Device: The Control Group

INTERVENTIONS:
Device: The Prism Adaptation Therapy Group — Once daily for a total of 20 sessions, in addition to the standard physical therapy and rehabilitation program, a pointing protocol was conducted under the supervision of the same physician/physiotherapist using prismatic-lens goggles.
  Arms: Prism Adaptation Therapy Group
Device: The Control Group — Once daily for a total of 20 sessions, in addition to the standard physical therapy and rehabilitation program, a pointing protocol was conducted under the supervision of the same physician/physiotherapist using neutral-lens goggles (sham goggles).
  Arms: Control Group

SUMMARY:
Complex Regional Pain Syndrome (CRPS) is a clinical condition characterized by pain that arises either without an identifiable triggering factor or with a severity disproportionate to the initiating event. Its progression is typically unpredictable, and most therapeutic interventions yield only partial efficacy. Prism Adaptation Therapy (PAT) is a sensorimotor training method traditionally employed to mitigate attentional deficits in post-stroke hemispatial neglect and has recently been explored as a treatment modality for CRPS. Preliminary non-blinded studies with small patient cohorts have demonstrated its potential to reduce pain and related symptoms. The present study aims to assess the effects of prism adaptation therapy administered during the acute phase on pain intensity and other clinical outcomes in CRPS, addressing the considerable challenges associated with managing chronic pain in this disorder.

DETAILED DESCRIPTION:
A total of 54 patients diagnosed with Complex Regional Pain Syndrome (CRPS) type 1, in accordance with the Budapest diagnostic criteria and fulfilling the inclusion and exclusion criteria, were enrolled in this study. Utilizing the sealed-envelope method, participants were randomized into two equal groups: 27 patients assigned to the prism adaptation therapy group and 27 to the control group. The control group received standard physical therapy and rehabilitation interventions supplemented by a pointing protocol administered once daily over 20 sessions under the supervision of the same physician/physiotherapist, with the use of neutral-lens goggles. Conversely, the prism adaptation therapy group underwent the identical pointing protocol employing prismatic-lens goggles in conjunction with standard physical therapy and rehabilitation interventions.

Baseline data collection prior to randomization included demographic characteristics such as age (years), sex (female/male), marital status (married/single), occupation, educational level, living arrangement, and alcohol and tobacco consumption. Clinical and disease-related baseline variables were also recorded, comprising height (cm), body weight (kg), body mass index (kg/m²), comorbidities, and current medication regimens. The etiology or inciting event(s) were documented, including fracture, surgery, immobilization, and casting. For fracture-related cases, detailed information on fracture pattern, intra-articular involvement, casting, surgical intervention, type and duration of immobilization, and the interval from the inciting event(s) to presentation at the physical medicine and rehabilitation outpatient clinic was noted. Furthermore, CRPS-associated signs and symptoms-including pain, edema, color changes, temperature alterations or asymmetry, sweating changes, nail and hair abnormalities, involuntary movements, tremor, weakness, and limitations in hand and wrist range of motion-were assessed at baseline. Sensory evaluations encompassed hyperalgesia testing with cotton wool and allodynia assessment using a 22-gauge black-tipped needle.

All patients were evaluated at three time points: baseline prior to treatment initiation (T0), immediately following treatment completion (T1), and six weeks post-treatment (T2). Assessments included clinical parameters, standardized evaluation tests, and ultrasonographic examinations.

ELIGIBILITY:
Inclusion Criteria

* Individuals aged between 18 and 75 years
* Patients diagnosed with CRPS Type 1 according to the IASP 2003 CRPS Budapest diagnostic criteria
* Presence of traumatic etiologies, including surgical procedures, fractures, or immobilization
* Patients who consented to participate and provided written informed consent

Exclusion Criteria

* History of inflammatory, autoimmune, hematologic, or neoplastic diseases
* Diabetes mellitus, thyroid disorders, hepatic or renal failure
* History of cranial trauma or cranial surgery within the preceding 6 months
* Use of diuretics, anti-inflammatory, antineoplastic, corticosteroid, immunosuppressive, antidepressant, or anxiolytic medications within the past 2 months
* Use of anticholinergic medications within the past 7 days
* Active ocular infection, inflammation, allergy, or recent use/exposure to ophthalmic drops
* History of lens or ocular surgery within the last 3 months
* Current or previous use of glasses or contact lenses, or diagnosis of refractive error ≥0.5 diopters
* Peripheral nerve injury in the affected hand consistent with CRPS Type 2 as per Budapest criteria
* Known progressive or non-progressive peripheral or central nervous system disorders
* CRPS Type 1 developing subsequent to central nervous system injury (e.g., stroke)
* Patients in the acute phase following primary or secondary tendon repair
* Presence of comorbid conditions likely to impair functionality and health-related quality of life, such as decompensated heart failure, chronic kidney failure, or malignancy
* Comorbid diseases affecting hand function, including rheumatoid arthritis, psoriatic arthritis, or other inflammatory disorders involving the hand
* Joint restriction and/or muscle weakness in the affected extremity that would impede movement
* History of acute upper-extremity deep vein thrombosis or arterial thrombosis
* Arterial or venous injury and/or history of arterial or venous repair surgery
* History of heavy alcohol consumption or inappropriate opioid use
* Inadequately treated psychiatric disorders or conditions, such as major depression, anxiety, or schizophrenia
* Recurrent diagnosis of CRPS Type 1, defined as patients experiencing repeated episodes

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2023-10-04 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | Baseline, post-treatment (Week 4), and follow-up (Week 10)
  The visual analog scale (VAS) is an instrument used to quantify pain intensity. It can be presented in either a vertical or horizontal orientation. Patients are asked, "If 10 represents the worst pain imaginable and 0 represents no pain, how much pain are you experiencing at this moment?" The scale consists of a 100-mm straight line on which patients indicate the severity of their symptoms. The left endpoint is typically labeled "no pain," while the right endpoint is labeled "worst pain imaginable." Patients mark the point on the line that best corresponds to their perceived pain level. The distance from the left endpoint to the marked point is then measured and recorded as the pain score.
LANNS | Baseline, post-treatment (Week 4), and follow-up (Week 10)
  The LANSS is employed to evaluate neuropathic pain. It comprises five pain-related questions and two sensory assessments.In the sensory assessment section, allodynia and pin-prick sensation are examined. A score of 12 or above indicates that the pain is likely neuropathic in nature. The maximum total score is 24.

SECONDARY OUTCOMES:
Evaluation of Joint Range of Motion | Baseline, post-treatment (Week 4), and follow-up (Week 10)
  Range of motion was assessed using a goniometer for the wrist (flexion/extension, radial/ulnar deviation) and the forearm (supination/pronation). Each measurement was performed three times, and the mean value was calculated and recorded.
Assessment of Light Touch Sensation | Baseline, post-treatment (Week 4), and follow-up (Week 10)
  Light touch sensation was evaluated using Semmes-Weinstein monofilaments (SWM). The assessment was conducted at seven sites corresponding to the dermatomal distribution of the median, radial, and ulnar nerves. During the procedure, patients were instructed to avert their gaze from the tested area. Each filament was applied perpendicularly for 1.5 seconds until it bent. Patients were asked to indicate when they perceived the stimulus. Filaments within the 1.65-4.08 range were applied three times, whereas those within the 4.17-6.65 range were applied once, and the patient's response was recorded. Values between 1.65 and 2.83 (green) were classified as normal; 3.22-3.61 (blue) indicated diminished light touch; 3.84-4.31 (purple) signified diminished protective sensation; and 4.56-6.65 (red) represented loss of protective sensation. In cases where there was no response to the 6.65 filament, this was documented as no response, and deep pressure sensation was subsequently assessed.
Assessment of Grip and Lateral Pinch Strength | Baseline, post-treatment (Week 4), and follow-up (Week 10)
  Grip strength and lateral pinch strength were assessed using a Lafayette digital hand dynamometer. Grip strength measurements were conducted in the seated position as recommended by the American Society of Hand Therapists (ASHT), with the wrist maintained in a neutral position, the forearm supported in mid-rotation, the elbow flexed at 90°, and the shoulder positioned neutrally with adduction. Each measurement was performed three times per patient, and the mean value was calculated.
  For lateral pinch strength, the dynamometer was pressed using the distal phalanx of the thumb, supported against the lateral aspect of the second phalanx of the index finger. Patients were instructed to exert maximal force during the measurement. Each measurement was repeated three times per patient, and the average value was recorded.
Measurement of Wrist Circumference | Baseline, post-treatment (Week 4), and follow-up (Week 10)
  Wrist circumference was measured in all patients using a measuring tape, carefully positioned to fit precisely over the styloid processes of the radius and ulna. To ensure measurement reliability, each assessment was conducted three times, and the mean value was recorded. Measurements were reported in centimeters.
Assessment of Hand and Wrist Volume | Baseline, post-treatment (Week 4), and follow-up (Week 10)
  The assessment of extremity volume is considered the gold standard for volumetric measurements. For each patient, the volumeter was filled with water until it overflowed, and the extremity to be measured was immersed such that the thumb faced the opening of the volumeter and the web space between the second and third fingers aligned with the marked midpoint of the volumeter. The volume of the displaced water was measured using a graduated container for both the healthy and affected extremities of each patient. Measurements were repeated three times separately, recorded individually, and the average value was determined in milliliters (ml).
Evaluation of Manual Dexterity | Baseline, post-treatment (Week 4), and follow-up (Week 10)
  Upper-extremity function was evaluated using the Nine-Hole Peg Test. Participants were instructed to sequentially pick up nine pegs from the side compartment, insert them one by one into the nine holes on the board, and then remove them as quickly as possible. The time taken to complete the task was recorded using a stopwatch. Completion times were standardized based on participants' age, sex, and dominant hand. The test was administered three times per participant, and the mean completion time was calculated.
Assessment of Functional Status in Activities of Daily Living (ADL) | Baseline, post-treatment (Week 4), and follow-up (Week 10)
  The hand function of the patients included in the study was assessed using the Duruöz Hand Index (DHI), an 18-item questionnaire that does not require prior training or specialized equipment. The questionnaire evaluates activities of daily living categorized into domains such as kitchen tasks, dressing, hygiene and cleaning, work-related activities, and other routine daily functions. Each item is scored on a Likert scale, resulting in a total score ranging from 0 to 90, where lower scores correspond to better functional ability.
Assessment of Disability | Baseline, post-treatment (Week 4), and follow-up (Week 10)
  Disability in all participants was evaluated using the Quick Disabilities of the Arm, Shoulder, and Hand (QuickDASH) questionnaire to assess limitations in activity and participation.
Assessment of Quality of Life | Baseline, post-treatment (Week 4), and follow-up (Week 10)
  To evaluate quality of life, all participants completed the Short Form-36 Health Survey (SF-36). Initially comprising 149 items in 1999, the instrument was subsequently refined to the SF-20. To expand the assessment's scope and improve its psychometric robustness, the 36-item version was developed. The SF-36 consists of 36 items categorized into eight subscales.
  Respondents are instructed to consider their experiences over the preceding four weeks. An alternative version assessing the prior one week is also available to capture acute changes. Items 4 and 5 are answered with binary (yes/no) responses, while the remaining items utilize Likert-type scales with three to six response options. Each subscale is scored independently on a scale from 0 to 100, where higher scores denote better health status.
Assessment of Kinesiophobia | Baseline, post-treatment (Week 4), and follow-up (Week 10)
  Patients were evaluated using the Tampa Scale for Kinesiophobia (TSK), a 17-item questionnaire designed to assess fear of movement and/or re-injury. The total score ranges from 17 (lowest) to 68 (highest), with elevated scores indicating greater kinesiophobia, which corresponds to an increased fear of movement and falling.
Ultrasonographic Assessment | Baseline, post-treatment (Week 4), and follow-up (Week 10)
  Ultrasonographic measurements of all patients included in the study were conducted using a G.E. LOGIQ P5 ultrasound system. The device frequency was set between 7 and 12 MHz, and measurements were obtained by positioning a linear transducer over the third metacarpophalangeal joint of the affected limb. Echogenicity, subcutaneous tissue structure, and edema characteristics were assessed, and the findings were classified according to the Ultrasonographic Subcutaneous Edema Grading (USEG) scale.

CONTACTS AND LOCATIONS:
Overall Officials: ECE ÜNLÜ AKYÜZ, MD, Prof., Study Director — Ankara Etlik City Hospital
Locations (1):
- Ankara Etlik City Hospital, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared publicly due to institutional policies and ethical considerations. De-identified, aggregate results will be reported in publications.